CLINICAL TRIAL: NCT04298229
Title: A Randomized, Open-label Study of Dapagliflozin in Patients With or Without Type 2 Diabetes Admitted With Acute Heart Failure
Brief Title: Efficacy and Safety of Dapagliflozin in Acute Heart Failure
Acronym: DICTATE-AHF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Zachary L. Cox, Co-Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200017
Record Dates: First submitted 2020-03-02; First posted 2020-03-06 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Participants will be recruited following an initial standard evaluation in the ED and randomized within 24 hours of presentation for ADHF in a 1:1 fashion to protocolized diuretic therapy or dapagliflozin + protocolized diuretic therapy.
Who Masked: Outcomes Assessor
Masking Description: The Clinical Event Adjudication Committee will consist of 3 independent clinicians, which will consist of at least one endocrinologist and at least one heart failure specialist. The members of this committee will be independent of the study implementation teams and will be blinded to study arm assignment. This committee will review abstracted clinical data to determine when primary endpoints and major events have occurred. The CEAC will review data for the following study outcomes:
  * Potential in-hospital worsening heart failure events
  * 30-day readmission events for heart failure or diabetes-related care
  * Prolonged hospitalization as a result of the following safety outcomes: hypotension requiring medical intervention or hypoglycemia requiring medical intervention
  * Inpatient mortality events
  * Potential ketoacidosis events
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Protocolized diuretic therapy (Active Comparator): The patients with diabetes will receive standard of care point of care blood glucose monitoring 4 times daily (before meals and at bedtime) and sliding scale insulin.
  The initial loop diuretic regimen after enrollment:
  Loop diuretic naïve: If the patient does not take a scheduled loop diuretic as an outpatient, the initial IV loop diuretic dose will be 40mg of furosemide equivalents every 12 hours.
  Chronic, oral loop diuretic therapy: If the patient takes a scheduled loop diuretic regimen as an outpatient prior to hospital admission, the initial IV loop diuretic daily dose will be 2 times the total daily home regimen dose. Diuretic therapy will be titrated to goal urine output using a standardized diuretic protocol.
  Interventions: Other: Protocolized Diuretic Therapy
- Protocolized diuretic therapy plus SGLT2 inhibitor therapy (Experimental): The patients with diabetes will receive standard of care point of care blood glucose monitoring 4 times daily (before meals and at bedtime) and sliding scale insulin.
  The initial loop diuretic regimen after enrollment:
  Loop diuretic naïve: If the patient does not take a scheduled loop diuretic as an outpatient, the initial IV loop diuretic dose will be 40mg of furosemide equivalents every 12 hours.
  Chronic, oral loop diuretic therapy: If the patient takes a scheduled loop diuretic regimen as an outpatient prior to hospital admission, the initial IV loop diuretic daily dose will be 2 times the total daily home regimen dose. Diuretic therapy will be titrated to goal urine output using a standardized diuretic protocol.
  The patient will receive SGLT2 inhibitor therapy with dapagliflozin 10 mg orally once daily until 5 days or hospital discharge.
  Interventions: Drug: Dapagliflozin 10 MG; Other: Protocolized Diuretic Therapy

INTERVENTIONS:
Drug: Dapagliflozin 10 MG — SGLT2 inhibitors being investigated for its diuretic and natriuretic effects on top of protocolized diuretic therapy.
  Other Names: sodium-glucose cotransporter-2(SGLT2) inhibitors
  Arms: Protocolized diuretic therapy plus SGLT2 inhibitor therapy
Other: Protocolized Diuretic Therapy — Structured usual care arm with protocolized diuretic therapy based on urine output.

SUMMARY:
This is a randomized trial of the addition of dapagliflozin to patients with or without type 2 diabetes hospitalized with acute decompensated heart failure (ADHF). Participants will be recruited following an initial standard evaluation in the ED and randomized within 24 hours of presentation for ADHF in a 1:1 fashion to protocolized diuretic therapy or dapagliflozin + protocolized diuretic therapy.

DETAILED DESCRIPTION:
Patients with acute decompensated HF (ADHF) are generally admitted due to symptoms of congestion and 90% are treated with a loop diuretic. However at least one-third of these patients are inadequately decongested due primarily to "diuretic resistance" and/ or "cardiorenal syndrome". The inability to achieve decongestion is associated with a worse prognosis and a higher rate of re-hospitalization for ADHF. More than 40% of all patients admitted with ADHF have diabetes and that percentage is growing both in Heart Failure with Reduced Ejection Fraction (HFrEF) and Preserved Ejection Fraction (HFpEF).

The admission blood glucose is elevated in approximately one-half of ADHF hospitalizations. We recently demonstrated the admission blood glucose was within 50mg/dl of the chronic average blood glucose in 66% of patients with diabetes admitted with ADHF. The median (IQR) admission blood glucose change from the chronic blood glucose was only -7 (-29, 26) mg/dl. Thus, the acute glucose in patients with T2DM presenting with acute heart failure is most often related to poor chronic glucose control suggesting that these patients would benefit from attempts to initiate therapies to improve chronic glucose control while in the hospital.

No new therapies have been introduced in the United States for ADHF in several decades. Natriuretic peptides such as nesiritide and ularitide have failed to improve outcomes in either the chronic or acute heart failure patients. Diuretic resistance and hyperglycemia are common problems in ADHF admissions and represent a therapeutic opportunity for new therapies.

The sodium-glucose cotransporter-2(SGLT2) inhibitors, now approved for the anti-hyperglycemic therapies also have an osmotic diuretic and natriuretic effect. In the chronic setting SGLT2 inhibitors reduce weight with modest decrements in systolic and diastolic blood pressure with a marked drop in albuminuria and a small drop in estimated GFR (-5 mL min-1.1.73 m-2) which returns to baseline over time. In patients with diabetes the SGLT2 transporter likely accounts for as much as 14% of total sodium chloride absorption. In the acute setting following a single dose, SGLT2 inhibitors did not increase urine volume. However, the acute diuretic effects have not been studied in a population with heart failure with or without concomitant hyperglycemia who are undergoing diuresis. To our knowledge, no current trials are investigating the effects of SGLT2 inhibition in ADHF. The current studies planned in HF are investigating the acute effects of SGLT2 on stable HF (NCT03027960), the chronic effects of SGLT2 inhibition in compensated, chronic HF (NCT03619213, NCT02653482, NCT03030235, NCT03057977), changes in pulmonary pressure hemodynamics in patients monitored by CardioMEMs devices (NCT03030222), and effects on cardiopulmonary exercise fitness in chronic HF (NCT02862067).

Congestion remains the major cause of hospital readmission for heart failure and an inpatient plan of care that allowed more effective decongestion would be rapidly and widely adopted by the medical community. Therefore, we propose to test the decongesting effects of the SGLT2 inhibitor dapagliflozin in patients with or without Type II diabetes admitted with an acute decompensation of chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Randomized within 24 of presentation during a hospital admission for hypervolemic decompensated heart failure defined as:

  * pulmonary artery catheterization with a pulmonary capillary wedge pressure greater than 19mmHg plus a systemic physical exam finding of hypervolemia (peripheral edema, ascites, or pulmonary edema on auscultation)
  * in the absence of pulmonary artery catheterization data 2 of the following signs or symptoms: peripheral edema, ascites, jugular venous pressure > 10mmHg, orthopnea, paroxysmal nocturnal dyspnea, 5-pound weight gain, or signs of congestion on chest x-ray or lung ultrasound
* Planned use of IV loop diuretic therapy during current hospitalization
* eGFR of 25 ml/min/1.73m2 by the MDRD equation or greater

Exclusion Criteria:

* Type 1 diabetes
* Serum glucose < 80mg/dl at enrollment
* Systolic blood pressure < 90mmHg at enrollment
* Requirement of intravenous inotropic therapy or anticipated need during the study
* History of hypersensitivity to any SGLT2 inhibitors
* Women who are pregnant or breastfeeding
* Severe anemia (Hemoglobin < 7.5g/dl)
* Severe uncorrected aortic or mitral stenosis
* Inability to perform standing weights or measure urine output accurately
* History of diabetic ketoacidosis
* Scheduled combination nephron blockade with loop and thiazide therapy as an outpatient for more than 7 days prior to admission (excluding HCTZ < 50mg for blood pressure)
* Diffuse anasarca with 4+ edema and projected hypervolemia exceeding 40-pounds
* Severe hepatic impairment (Child-Pugh class C)
* Clinical picture consistent with acute myocardial infarction including troponin rise and fall or ischemic changes on electrocardiogram
* Site investigator determines the subject is not a good candidate to participate in the study at this tine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn Lindenfeld, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (6):
- United States (6):
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of North Carolina, Chapel Hill, North Carolina
  - INTEGRIS, Oklahoma City, Oklahoma
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - Saint Thomas West Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams KF Jr, Fonarow GC, Emerman CL, LeJemtel TH, Costanzo MR, Abraham WT, Berkowitz RL, Galvao M, Horton DP; ADHERE Scientific Advisory Committee and Investigators. Characteristics and outcomes of patients hospitalized for heart failure in the United States: rationale, design, and preliminary observations from the first 100,000 cases in the Acute Decompensated Heart Failure National Registry (ADHERE). Am Heart J. 2005 Feb;149(2):209-16. doi: 10.1016/j.ahj.2004.08.005. PMID 15846257
- [Background] Chioncel O, Mebazaa A, Maggioni AP, Harjola VP, Rosano G, Laroche C, Piepoli MF, Crespo-Leiro MG, Lainscak M, Ponikowski P, Filippatos G, Ruschitzka F, Seferovic P, Coats AJS, Lund LH; ESC-EORP-HFA Heart Failure Long-Term Registry Investigators. Acute heart failure congestion and perfusion status - impact of the clinical classification on in-hospital and long-term outcomes; insights from the ESC-EORP-HFA Heart Failure Long-Term Registry. Eur J Heart Fail. 2019 Nov;21(11):1338-1352. doi: 10.1002/ejhf.1492. Epub 2019 May 24. PMID 31127678
- [Background] Damman K, Testani JM. The kidney in heart failure: an update. Eur Heart J. 2015 Jun 14;36(23):1437-44. doi: 10.1093/eurheartj/ehv010. Epub 2015 Apr 2. PMID 25838436
- [Background] Echouffo-Tcheugui JB, Xu H, DeVore AD, Schulte PJ, Butler J, Yancy CW, Bhatt DL, Hernandez AF, Heidenreich PA, Fonarow GC. Temporal trends and factors associated with diabetes mellitus among patients hospitalized with heart failure: Findings from Get With The Guidelines-Heart Failure registry. Am Heart J. 2016 Dec;182:9-20. doi: 10.1016/j.ahj.2016.07.025. Epub 2016 Aug 27. PMID 27914505
- [Background] Mebazaa A, Gayat E, Lassus J, Meas T, Mueller C, Maggioni A, Peacock F, Spinar J, Harjola VP, van Kimmenade R, Pathak A, Mueller T, Tavazzi L, Disomma S, Metra M, Pascual-Figal D, Laribi S, Logeart D, Nouira S, Sato N, Parenica J, Deye N, Boukef R, Collet C, Van den Berghe G, Cohen-Solal A, Januzzi JL Jr; GREAT Network. Association between elevated blood glucose and outcome in acute heart failure: results from an international observational cohort. J Am Coll Cardiol. 2013 Feb 26;61(8):820-9. doi: 10.1016/j.jacc.2012.11.054. Epub 2013 Jan 16. PMID 23333145
- [Background] Kosiborod M, Inzucchi SE, Spertus JA, Wang Y, Masoudi FA, Havranek EP, Krumholz HM. Elevated admission glucose and mortality in elderly patients hospitalized with heart failure. Circulation. 2009 Apr 14;119(14):1899-907. doi: 10.1161/CIRCULATIONAHA.108.821843. Epub 2009 Mar 30. PMID 19332465
- [Background] Cox ZL, Lai P, Lewis CM, Lindenfeld J. Change in admission blood glucose from chronic glycemic status in acute heart failure hospitalization and 30-day outcomes: A retrospective analysis. Int J Cardiol. 2020 Jan 15;299:180-185. doi: 10.1016/j.ijcard.2019.07.069. Epub 2019 Jul 23. PMID 31395364
- [Background] Packer M, O'Connor C, McMurray JJV, Wittes J, Abraham WT, Anker SD, Dickstein K, Filippatos G, Holcomb R, Krum H, Maggioni AP, Mebazaa A, Peacock WF, Petrie MC, Ponikowski P, Ruschitzka F, van Veldhuisen DJ, Kowarski LS, Schactman M, Holzmeister J; TRUE-AHF Investigators. Effect of Ularitide on Cardiovascular Mortality in Acute Heart Failure. N Engl J Med. 2017 May 18;376(20):1956-1964. doi: 10.1056/NEJMoa1601895. Epub 2017 Apr 12. PMID 28402745
- [Background] O'Connor CM, Starling RC, Hernandez AF, Armstrong PW, Dickstein K, Hasselblad V, Heizer GM, Komajda M, Massie BM, McMurray JJ, Nieminen MS, Reist CJ, Rouleau JL, Swedberg K, Adams KF Jr, Anker SD, Atar D, Battler A, Botero R, Bohidar NR, Butler J, Clausell N, Corbalan R, Costanzo MR, Dahlstrom U, Deckelbaum LI, Diaz R, Dunlap ME, Ezekowitz JA, Feldman D, Felker GM, Fonarow GC, Gennevois D, Gottlieb SS, Hill JA, Hollander JE, Howlett JG, Hudson MP, Kociol RD, Krum H, Laucevicius A, Levy WC, Mendez GF, Metra M, Mittal S, Oh BH, Pereira NL, Ponikowski P, Tang WH, Tanomsup S, Teerlink JR, Triposkiadis F, Troughton RW, Voors AA, Whellan DJ, Zannad F, Califf RM. Effect of nesiritide in patients with acute decompensated heart failure. N Engl J Med. 2011 Jul 7;365(1):32-43. doi: 10.1056/NEJMoa1100171. PMID 21732835
- [Background] Cox ZL, Lenihan DJ. Loop diuretic resistance in heart failure: resistance etiology-based strategies to restoring diuretic efficacy. J Card Fail. 2014 Aug;20(8):611-22. doi: 10.1016/j.cardfail.2014.05.007. Epub 2014 May 28. PMID 24879974
- [Background] Heerspink HJ, Perkins BA, Fitchett DH, Husain M, Cherney DZ. Sodium Glucose Cotransporter 2 Inhibitors in the Treatment of Diabetes Mellitus: Cardiovascular and Kidney Effects, Potential Mechanisms, and Clinical Applications. Circulation. 2016 Sep 6;134(10):752-72. doi: 10.1161/CIRCULATIONAHA.116.021887. Epub 2016 Jul 28. PMID 27470878
- [Background] Heise T, Seewaldt-Becker E, Macha S, Hantel S, Pinnetti S, Seman L, Woerle HJ. Safety, tolerability, pharmacokinetics and pharmacodynamics following 4 weeks' treatment with empagliflozin once daily in patients with type 2 diabetes. Diabetes Obes Metab. 2013 Jul;15(7):613-21. doi: 10.1111/dom.12073. Epub 2013 Feb 17. PMID 23356556
- [Background] Testani JM, Brisco MA, Turner JM, Spatz ES, Bellumkonda L, Parikh CR, Tang WH. Loop diuretic efficiency: a metric of diuretic responsiveness with prognostic importance in acute decompensated heart failure. Circ Heart Fail. 2014 Mar 1;7(2):261-70. doi: 10.1161/CIRCHEARTFAILURE.113.000895. Epub 2013 Dec 30. PMID 24379278
- [Background] Palazzuoli A, Testani JM, Ruocco G, Pellegrini M, Ronco C, Nuti R. Different diuretic dose and response in acute decompensated heart failure: Clinical characteristics and prognostic significance. Int J Cardiol. 2016 Dec 1;224:213-219. doi: 10.1016/j.ijcard.2016.09.005. Epub 2016 Sep 10. PMID 27657476
- [Background] Lala A, McNulty SE, Mentz RJ, Dunlay SM, Vader JM, AbouEzzeddine OF, DeVore AD, Khazanie P, Redfield MM, Goldsmith SR, Bart BA, Anstrom KJ, Felker GM, Hernandez AF, Stevenson LW. Relief and Recurrence of Congestion During and After Hospitalization for Acute Heart Failure: Insights From Diuretic Optimization Strategy Evaluation in Acute Decompensated Heart Failure (DOSE-AHF) and Cardiorenal Rescue Study in Acute Decompensated Heart Failure (CARESS-HF). Circ Heart Fail. 2015 Jul;8(4):741-8. doi: 10.1161/CIRCHEARTFAILURE.114.001957. Epub 2015 Jun 3. PMID 26041600
- [Background] Kronmal RA. Spurious Correlation and the Fallacy of the Ratio Standard Revisited. J Roy Stat Soc a Sta. 1993;156:379-392.
- [Background] Walker SH, Duncan DB. Estimation of the probability of an event as a function of several independent variables. Biometrika. 1967 Jun;54(1):167-79. No abstract available. PMID 6049533
- [Background] Harrell FE. Regression Modeling Strategies: With Applications to Linear Models, Logistic and Ordinal Regression, and Survival Analysis, 2nd Edition. Springer Ser Stat. 2015.
- [Background] Teerlink JR, Cotter G, Davison BA, Felker GM, Filippatos G, Greenberg BH, Ponikowski P, Unemori E, Voors AA, Adams KF Jr, Dorobantu MI, Grinfeld LR, Jondeau G, Marmor A, Masip J, Pang PS, Werdan K, Teichman SL, Trapani A, Bush CA, Saini R, Schumacher C, Severin TM, Metra M; RELAXin in Acute Heart Failure (RELAX-AHF) Investigators. Serelaxin, recombinant human relaxin-2, for treatment of acute heart failure (RELAX-AHF): a randomised, placebo-controlled trial. Lancet. 2013 Jan 5;381(9860):29-39. doi: 10.1016/S0140-6736(12)61855-8. Epub 2012 Nov 7. PMID 23141816
- [Background] Konstam MA, Gheorghiade M, Burnett JC Jr, Grinfeld L, Maggioni AP, Swedberg K, Udelson JE, Zannad F, Cook T, Ouyang J, Zimmer C, Orlandi C; Efficacy of Vasopressin Antagonism in Heart Failure Outcome Study With Tolvaptan (EVEREST) Investigators. Effects of oral tolvaptan in patients hospitalized for worsening heart failure: the EVEREST Outcome Trial. JAMA. 2007 Mar 28;297(12):1319-31. doi: 10.1001/jama.297.12.1319. Epub 2007 Mar 25. PMID 17384437
- [Background] Felker GM, Mentz RJ, Cole RT, Adams KF, Egnaczyk GF, Fiuzat M, Patel CB, Echols M, Khouri MG, Tauras JM, Gupta D, Monds P, Roberts R, O'Connor CM. Efficacy and Safety of Tolvaptan in Patients Hospitalized With Acute Heart Failure. J Am Coll Cardiol. 2017 Mar 21;69(11):1399-1406. doi: 10.1016/j.jacc.2016.09.004. Epub 2016 Sep 18. PMID 27654854
- [Background] Konstam MA, Kiernan M, Chandler A, Dhingra R, Mody FV, Eisen H, Haught WH, Wagoner L, Gupta D, Patten R, Gordon P, Korr K, Fileccia R, Pressler SJ, Gregory D, Wedge P, Dowling D, Romeling M, Konstam JM, Massaro JM, Udelson JE; SECRET of CHF Investigators, Coordinators, and Committee Members. Short-Term Effects of Tolvaptan in Patients With Acute Heart Failure and Volume Overload. J Am Coll Cardiol. 2017 Mar 21;69(11):1409-1419. doi: 10.1016/j.jacc.2016.12.035. PMID 28302292
- [Background] Chen HH, Anstrom KJ, Givertz MM, Stevenson LW, Semigran MJ, Goldsmith SR, Bart BA, Bull DA, Stehlik J, LeWinter MM, Konstam MA, Huggins GS, Rouleau JL, O'Meara E, Tang WH, Starling RC, Butler J, Deswal A, Felker GM, O'Connor CM, Bonita RE, Margulies KB, Cappola TP, Ofili EO, Mann DL, Davila-Roman VG, McNulty SE, Borlaug BA, Velazquez EJ, Lee KL, Shah MR, Hernandez AF, Braunwald E, Redfield MM; NHLBI Heart Failure Clinical Research Network. Low-dose dopamine or low-dose nesiritide in acute heart failure with renal dysfunction: the ROSE acute heart failure randomized trial. JAMA. 2013 Dec 18;310(23):2533-43. doi: 10.1001/jama.2013.282190. PMID 24247300
- [Background] Voors AA, Davison BA, Teerlink JR, Felker GM, Cotter G, Filippatos G, Greenberg BH, Pang PS, Levin B, Hua TA, Severin T, Ponikowski P, Metra M; RELAX-AHF Investigators. Diuretic response in patients with acute decompensated heart failure: characteristics and clinical outcome--an analysis from RELAX-AHF. Eur J Heart Fail. 2014 Nov;16(11):1230-40. doi: 10.1002/ejhf.170. Epub 2014 Oct 7. PMID 25287144
- [Background] ter Maaten JM, Dunning AM, Valente MA, Damman K, Ezekowitz JA, Califf RM, Starling RC, van der Meer P, O'Connor CM, Schulte PJ, Testani JM, Hernandez AF, Tang WH, Voors AA. Diuretic response in acute heart failure-an analysis from ASCEND-HF. Am Heart J. 2015 Aug;170(2):313-21. doi: 10.1016/j.ahj.2015.05.003. Epub 2015 May 9. PMID 26299229
- [Background] Valente MA, Voors AA, Damman K, Van Veldhuisen DJ, Massie BM, O'Connor CM, Metra M, Ponikowski P, Teerlink JR, Cotter G, Davison B, Cleland JG, Givertz MM, Bloomfield DM, Fiuzat M, Dittrich HC, Hillege HL. Diuretic response in acute heart failure: clinical characteristics and prognostic significance. Eur Heart J. 2014 May 14;35(19):1284-93. doi: 10.1093/eurheartj/ehu065. Epub 2014 Feb 28. PMID 24585267
- [Background] Ter Maaten JM, Valente MA, Damman K, Cleland JG, Givertz MM, Metra M, O'Connor CM, Teerlink JR, Ponikowski P, Bloomfield DM, Cotter G, Davison B, Subacius H, van Veldhuisen DJ, van der Meer P, Hillege HL, Gheorghiade M, Voors AA. Combining Diuretic Response and Hemoconcentration to Predict Rehospitalization After Admission for Acute Heart Failure. Circ Heart Fail. 2016 Jun;9(6):e002845. doi: 10.1161/CIRCHEARTFAILURE.115.002845. PMID 27266853
- [Derived] Cox ZL, Collins SP, Hernandez GA, McRae AT 3rd, Davidson BT, Adams K, Aaron M, Cunningham L, Jenkins CA, Lindsell CJ, Harrell FE Jr, Kampe C, Miller KF, Stubblefield WB, Lindenfeld J. Efficacy and Safety of Dapagliflozin in Patients With Acute Heart Failure. J Am Coll Cardiol. 2024 Apr 9;83(14):1295-1306. doi: 10.1016/j.jacc.2024.02.009. PMID 38569758

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 240 patients were randomized to either Structured usual care or Dapagliflozin plus Structured usual care treatment arms
Groups:
- Structured Usual Care: Protocolized Diuretic Therapy: Structured usual care arm with protocolized diuretic therapy based on urine output.
- Dapagliflozin Plus Structured Usual Care: Dapagliflozin 10 MG: SGLT2 inhibitors being investigated for its diuretic and natriuretic effects on top of protocolized diuretic therapy.
  Protocolized Diuretic Therapy: Structured usual care arm with protocolized diuretic therapy based on urine output.
Period: Overall Study
Arm/Group | Structured Usual Care | Dapagliflozin Plus Structured Usual Care
Started | 120 | 120
Completed | 116 | 118
Not Completed | 4 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Did not receive IV loop diuretics | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Structured Usual Care: Structured usual care arm with protocolized diuretic therapy based on urine output.
- Dapagliflozin + Structured Usual Care: Dapagliflozin 10 MG once daily + Structured usual care arm with protocolized diuretic therapy based on urine output.
- Total: Total of all reporting groups
Arm/Group | Structured Usual Care | Dapagliflozin + Structured Usual Care | Total
Number analyzed (Participants) | 119 | 119 | 238
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [55 to 74] | 65 [56 to 73] | 65 [56 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 41 | 93
  Male | 67 | 78 | 145
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 39 | 68
  White | 84 | 79 | 163
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 1 | 7
Left ventricular ejection fraction [Median (Inter-Quartile Range); unit: Percentage of ejection fraction] | 35 [25 to 60] | 45 [26 to 56] | 40 [25 to 60]
systolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 120 [110 to 136] | 121 [112 to 136] | 121 [110 to 136]
estimated Glomerular Filtration Rate (eGFR) [Median (Inter-Quartile Range); unit: mL/min/1.73m2] | 54 [40 to 71] | 51 [43 to 68] | 53 [42 to 70]

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Change in Weight (Kilograms) Per 40mg of IV Furosemide Equivalents, Adjusted for Baseline Weight
Description: cumulative change in weight (kilograms) per 40mg of IV furosemide equivalents from enrollment to day 5 or discharge (if earlier) between protocolized diuretic therapy and dapagliflozin plus protocolized diuretic therapy guided by urine output
Time Frame: Baseline to Day 5 or discharge if earlier
Measure: Median (Inter-Quartile Range); unit: kg/40mg IV furosemide
Arm/Group | Structured Usual Care | Dapagliflozin Plus Structured Usual Care
Number analyzed (Participants) | 116 | 118
kg/40mg IV furosemide | -0.31 [-0.39 to -0.23] | -0.42 [-0.52 to -0.33]

2. Secondary Outcome: Number of Participants With Inpatient Worsening Heart Failure
Description: Number of participants with worsening heart failure during hospitalization requiring IV inotropic therapy with dobutamine, milrinone, or dopamine or admission to an intensive care unit as adjudicated by the Clinical Event Adjudication Committee
Time Frame: Baseline to hospital discharge, an average of 5 days
Measure: Number; unit: participants
Arm/Group | Structured Usual Care | Dapagliflozin + Structured Usual Care
Number analyzed (Participants) | 116 | 118
participants | 3 | 4

3. Secondary Outcome: Hospital Readmission
Description: Hospital readmission within 30 days of discharge for heart failure or diabetic reasons as adjudicated by the Clinical Event Adjudication Committee
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Structured Usual Care | Dapagliflozin + Structured Usual Care
Number analyzed (Participants) | 116 | 118
Participants | 20 | 19

ADVERSE EVENTS:
Time Frame: Adverse events were assessment from enrollment through 30-days after hospital discharge, on average 36 days from baseline
Description: AE were collected during daily monitoring while the patient was hospitalized during the index hospitalization and via 30-day follow-up phone calls after discharge
Arm/Group | Structured Usual Care | Dapagliflozin + Structured Usual Care
All-Cause Mortality (participants affected / at risk) | 5/119 | 3/119
Serious Adverse Events (participants affected / at risk) | 7/119 | 6/119
Other Adverse Events (participants affected / at risk) | 17/119 | 13/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Structured Usual Care (N=119) | Dapagliflozin + Structured Usual Care (N=119)
Ketoacidosis (Endocrine disorders) | 0 (0) | 0 (0) — Ketoacidosis during the study period
Severe Hypotension (Cardiac disorders) | 1 (1) | 1 (1) — Hypotension prolonging hospitalization
Severe hypoglycemia (Endocrine disorders) | 0 (0) | 0 (0) — Hypoglycemia prolonging hospitalization
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 2 (2) — Stage 3 AKI using Acute Kidney Injury Network definition
Death (Cardiac disorders) | 5 (5) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Structured Usual Care (N=119) | Dapagliflozin + Structured Usual Care (N=119)
Hypoglycemia (Endocrine disorders) | 9 (9) | 7 (7)
HF exacerbation (Cardiac disorders) | 8 (8) | 6 (6) — Post-discharge worsening HF

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT04298229/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT04298229/SAP_001.pdf